CLINICAL TRIAL: NCT06336655
Title: Physiology of Unloading VA ECMO Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Principal Investigator, Joseph Tonna, Associate Professor, Division of Cardiothoracic Surgery, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 153309
Record Dates: First submitted 2024-03-08; First posted 2024-03-29 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-11

CONDITIONS: Cardiogenic Shock
Keywords: cardiogenic shock; extracorporeal membrane oxygenation; left ventricular unloading
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- With LV Unloading (Experimental): Patients on VA ECMO who randomize to receive LV unloading
  Interventions: Device: IABP
- Without LV Unloading (No Intervention): Patients on VA ECMO who randomize to receive no LV unloading

INTERVENTIONS:
Device: IABP — LV unloading via intra-aortic balloon pump (IABP)
  Other Names: LV unloading
  Arms: With LV Unloading

SUMMARY:
The goal of this clinical trial is to compare the use of veno-arterial extracorporeal membrane oxygenation (VA ECMO) with and without left ventricular (LV) unloading in patients being treated for cardiogenic shock (CS). The main aims of the study are:

1. To determine the physiologic effects on cardiopulmonary congestion of adding LV unloading to VA ECMO
2. To determine the effects on myocardial function of adding LV unloading to ECMO
3. To test the effects on myocardial recovery of adding LV unloading to VA ECMO

Participants who are being treated with VA ECMO will be randomized to receive or not receive LV unloading in the form of an intra-aortic balloon pump (IABP). Over the course of the study, the investigators will obtain measurements via lab work, echocardiography, and pulmonary artery catheter that will allow comparison of the two groups.

DETAILED DESCRIPTION:
Although extracorporeal membrane oxygenation (ECMO) for cardiogenic shock (CS) is used in over 3,000 patients per year, the best management strategies are not known. Identifying and improving treatment of CS is critically important, as CS occurs in 160,000 patients per year in the US with a 50% mortality rate. VA ECMO is an increasingly used method of mechanical circulatory support (MCS) for patients with CS refractory to medical therapy. Despite the benefit of full cardiopulmonary support ECMO is also thought to increase after load in the failing heart- which paradoxically reduces cardiac output and may lead to myocardial injury and cardiac congestion. A potential solution is to add a device to VA ECMO that decreases after-load - known as left ventricular (LV) unloading. LV unloading can be achieved with different approaches, directly with transvalvular pumps (known as a peripheral ventricular assist device (pVAD)), or indirectly with an intra-aortic balloon pump (IABP)

Preliminary data suggests that unloading the LV is associated with improved survival. Results from a cohort of VA ECMO patients with medical CS, showed a hospital survival benefit LV unloading (aOR 0.87 (0.79, 094); p=0.001). Data has also shown that the survival benefit of LV unloading was much larger with pVAD (HR 0.6), but with higher complications, including limb ischemia - a potentially catastrophic complication. However, results also show that different unloading approaches have different physiologic effects on the myocardium and on peripheral perfusion - highlighting the uncomfortable observation that it is not known how (physiologically) these unloading devices lead to changes in survival.

There are two potential pathways whereby LV unloading could influence survival, including myocardial effects (distension, injury, ejection fraction ) and peripheral effects (peripheral pulse pressure, lactate clearance, CO2 gap). Determining the physiologic effects from LV unloading according to device type and patient etiology will allow us to match the intervention with the patient's physiology. Data suggests that ECMO patients with acute myocardial infarction (AMI) have different mortality and different physiologic changes than patients with decompensated chronic heart failure (CHF) when unloaded.

The ultimate goal is to reduce morbidity and mortality in cardiogenic shock. This study will define the physiologic benefit of LV unloading during CS.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age 18 years or older)
* Diagnosis of acute cardiogenic shock (CS)
* Patients failing medical therapy, defined as 1 or more of the following:

  1. Society for Coronary Angiography and Interventions (SCAI) Stage C or greater
  2. 2 or more inotropic medications and not improving
  3. IABP in place and clinically worsening
  4. Placed on VA ECMO for CS
  5. In the opinion of the attending physician, patient has worsening CS and could require VA ECMO support in the near-term

Exclusion Criteria:

* Metastatic or stage 4 cancer
* Atrial septostomy
* Planned LV unloading on ECMO
* Anticipated death <72 hours
* Existing durable left ventricular assist device (dLVAD)
* Unwillingness to randomize
* Patients who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in pulmonary capillary wedge pressure | ECMO start, ECMO day 5, ECMO decannulation up to 3 months, day of ICU discharge up to 6 months
  Change in pulmonary capillary wedge pressure (PCWP) from ECMO start to ECMO day 5 (Day 5 - Baseline) with and without LV unloading

SECONDARY OUTCOMES:
Change in pulmonary artery diastolic pressure | ECMO start, ECMO days 1-5, ECMO decannulation up to 3 months, day of ICU discharge up to 6 months
  Change in pulmonary artery diastolic pressure (PADP) from ECMO start to ECMO day 5 (Day 5 - baseline) with and without LV unloading
Change in left ventricular end diastolic diameter | ECMO start, ECMO day 5, ECMO decannulation up to 3 months, day of ICU discharge up to 6 months
  Change in left ventricular end diastolic diameter (LVEDd) from ECMO start to ECMO day 5 (Day 5 - baseline) with and without LV unloading
Change in N-terminal pro b-type natriuretic peptide | ECMO start, ECMO days 1-5, ECMO decannulation up to 3 months, day of ICU discharge up to 6 months
  Change in N-terminal pro b-type natriuretic peptide (NT-pro BNP) from ECMO start to ECMO day 5 (Day 5 - baseline) with and without LV unloading
Hemodynamic stability | ECMO start, ECMO day 5
  Hemodynamic stability (defined as a change in mean arterial pressure [MAP] from prior to turn down until 2 minutes of wean) at ECMO day 5 with and without LV unloading
Global cardiovascular function | ECMO start, ECMO days 1-5
  Global cardiovascular function is defined as arterial pulse pressure during the protocoled wean. To assess this outcome, the investigators will calculate the change in pulse pressure from prior to wean to 2 minutes during wean.
Difference in partial pressure of carbon dioxide (pCO2) | ECMO start, q12 hours ECMO days 1-3, ECMO decannulation up to 3 months, day of ICU discharge up to 6 months
  As part of assessing global cardiovascular function, the investigators will measure, via lab draw, pCO2, which is the difference in CO2 between arterial and central venous blood. This is a marker of peripheral perfusion.
Lactate | ECMO start, ECMO days 1-5, ECMO decannulation up to 3 months, day of ICU discharge up to 6 months
  As part of assessing global cardiovascular function, the investigators will measure, via lab draw, arterial lactate. This is a marker of peripheral perfusion.
Cardiac BIN1 | ECMO start, ECMO day 5, day of ICU discharge up to 6 months
  Change in Cardiac BIN1 (cBIN1) serum level from Baseline to Day 5 (Day 5 - Baseline). cBIN1is a validated marker of myocardial recovery in heart failure.
Troponin I | ECMO start, ECMO days 1-5, ECMO decannulation up to 3 months, day of ICU discharge up to 6 months
  Change in troponin I from ECMO start to ECMO day 5 (Day 5 - Baseline)
Tumor necrosis factor alpha | ECMO start, ECMO day 5, ECMO decannulation up to 3 months, day of ICU discharge up to 6 months
  Change in tumor necrosis factor alpha (TNFa) from ECMO start to ECMO day 5 (Day 5 - Baseline)
Ejection fraction percentage | ECMO start, ECMO day 5, ECMO decannulation up to 3 months, day of ICU discharge up to 6 months
  Assessment of heart function via echocardiography
Interferon gamma | ECMO start, ECMO day 5, ECMO decannulation up to 3 months, day of ICU discharge up to 6 months
  Predictor of myocardial recovery assessed from baseline through ICU discharge
Limb ischemia | Randomization, 48 hours post-device removal
  Ischemia in the ipsilateral limb as the IABP will be tracked from baseline until 48 hours after the intervention is removed.
Mortality | Hospital discharge up to 6 months
  Assessment of patient mortality status at hospital discharge

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No